CLINICAL TRIAL: NCT01427608
Title: Sustaining Remission of Psychotic Depression
Acronym: STOP-PD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: University of Toronto (Other); University of Massachusetts, Worcester (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STOP-PD-II
Record Dates: First submitted 2011-08-30; First posted 2011-09-01 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Psychotic Depression
MeSH Terms: interventions — Sertraline; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline + Olanzapine (Active Comparator): Randomized to continue with sertraline and olanzapine under double-blind conditions.
  Interventions: Drug: Sertraline + Olanzapine
- Sertraline + Placebo (Placebo Comparator): Randomized to continue with sertraline and substitute placebo for olanzapine under double-blind conditions.
  Interventions: Drug: Sertraline + Placebo

INTERVENTIONS:
Drug: Sertraline + Olanzapine — Olanzapine 15mg/day. Adjustment of dose to 5mg/day to a maximum of 20mg/day will be permitted if necessitated by significant side-effects or clinical worsening
  Other Names: Zyprexa
  Arms: Sertraline + Olanzapine
Drug: Sertraline + Placebo — Taper from current dose of olanzapine to placebo over 4 weeks. Continue placebo for remainder of 36 week study.
  Other Names: Placebo
  Arms: Sertraline + Placebo

SUMMARY:
The acute phase of this study will monitor the response to a combination of an atypical antipsychotic medication olanzapine with an antidepressant medication sertraline in the acute treatment of the disorder. It is predicted that this combination will improve symptoms of psychotic depression and be associated metabolic side effects. Factors that moderate tolerability will be monitored. Improvement in symptoms could take between 4 and 12 weeks, followed by a period of 8 weeks during which participants will continue to take the same medications to stabilize the remission from symptoms of psychotic depression.

The maintenance phase will be a randomized, double-blind, placebo-controlled study of olanzapine for a period of up to 36 weeks to test whether continuing this combination decreases the risk of relapse and whether discontinuing the combination leads to improvement in metabolic measures. Subjects who complete the acute phase will be asked to consent separately to the randomized maintenance phase.

DETAILED DESCRIPTION:
The original STOP-PD study established that the combination of olanzapine and sertraline was significantly better than olanzapine alone in achieving remission of psychotic depression. This STOP-PD-II Sustaining Remission study aims to assess the long-term tolerability of taking this combination of medications and their efficacy at preventing a relapse of the symptoms. The acute phase of the study will monitor the efficacy and tolerability of the olanzapine and sertraline combination, including investigation of weight and metabolic variables, age effects on treatment response and tolerability, and the association of genetic polymorphisms to response or relapse. When subjects are stabilized on these medications for a period of 8 weeks they will be invited to participate in the randomized phase of the research: the olanzapine will be placebo-controlled, meaning half of the subjects will continue to take the olanzapine/sertraline combination and half will take a sertraline/placebo combination, for a period of 36 weeks. Symptoms and side effects will be monitored regularly throughout this phase. Randomization will be stratified on a 1:1 basis by age 60 and above.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-85 years, inclusive
2. Diagnosis: Diagnostic Statistical Manual-IV Trade Revision (DSM IV-TR) non-bipolar major depression with psychotic features established by both clinical interview with research psychiatrist and administration of SCID-IV.
3. Score >2 on Schedule for Affective Disorders (SADS) delusion severity item
4. Score >1 on any of the three conviction items of the Delusion Assessment Scale (DAS) (does not alter belief in response to reality testing)
5. 17-item HAM-D score of >20

Exclusion Criteria:

1. Current or lifetime DSM-IV-TR history of schizophrenia or other psychotic disorders or meeting current criteria for brief psychotic disorder, body dysmorphic disorder or obsessive-compulsive disorder
2. Current or lifetime DSM-IV-TR bipolar affective disorder
3. History of DSM-IV-TR defined alcohol or substance abuse or dependence within the past three months
4. Dementia or clinically significant cognitive impairment prior to index episode of depression, and/or a mean score >3 on 26-item caregiver assessment
5. Type 1 diabetes mellitus (defined as insulin-dependent diabetes mellitus with onset before age 35, and/or diabetes mellitus complicated by prior documented episode of ketoacidosis
6. Acute or unstable medical illness within the past 3 months; current abnormal serum free T4; current abnormally low vitamin B4 or folic acid level; medical conditions and/or medications for which psychotic or depressive symptoms can be a direct manifestation; neurological disease associated with extrapyramidal signs and symptoms; epilepsy, if the person has had one or more grand mal seizures within the past 12 months.
7. The need for treatment with any psychotropic medication other than sertraline, olanzapine or lorazepam; or with an anticonvulsant medication with mood-stabilizing properties.
8. Current pregnancy or plan to become pregnant during the course of the study; breast feeding in women with infants.
9. A documented history of being unable to tolerate olanzapine or sertraline including significant bradycardia (heart rate of <50 bpm), and serum sodium level of 129mmol/L or below.
10. History of non-response of the index episode of psychotic depression to at least a 6-week trial of at least 150mg/day sertraline combined with 15mg/day olanzapine
11. Patients showing ongoing improvement in current episode of psychotic depression with treatment other than sertraline or olanzapine
12. Patients who are in immediate need of electroconvulsive therapy (ECT) (imminent risk of suicide, refusing to eat, catatonic)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2011-10; Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Alexopoulos, MD, Principal Investigator — Weill Medical College of Cornell University; Alastair Flint, MD, Principal Investigator — University of Toronto; Anthony Rothschild, MD, Principal Investigator — University of Massachusetts, Worcester; Ellen Whyte, MD, Principal Investigator — University of Pittsburgh
Locations (4):
- United States (3):
  - Anthony Rothschild, MD, Worcester, Massachusetts
  - George Alexopoulos, MD, White Plains, New York
  - Ellen Whyte, MD, Pittsburgh, Pennsylvania
- Alastair Flint, MD, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neufeld NH, Oliver LD, Mulsant BH, Alexopoulos GS, Hoptman MJ, Tani H, Marino P, Meyers BS, Rothschild AJ, Whyte EM, Bingham KS, Flint AJ, Voineskos AN. Effects of antipsychotic medication on functional connectivity in major depressive disorder with psychotic features. Mol Psychiatry. 2023 Aug;28(8):3305-3313. doi: 10.1038/s41380-023-02118-8. Epub 2023 May 31. PMID 37258617
- [Derived] Bingham KS, Calarco N, Dickie EW, Alexopoulos GS, Butters MA, Meyers BS, Marino P, Neufeld NH, Rothschild AJ, Whyte EM, Mulsant BH, Flint AJ, Voineskos AN. The relationship of white matter microstructure with psychomotor disturbance and relapse in remitted psychotic depression. J Affect Disord. 2023 Aug 1;334:317-324. doi: 10.1016/j.jad.2023.04.136. Epub 2023 May 4. PMID 37149056
- [Derived] Flint AJ, Bingham KS, Alexopoulos GS, Marino P, Mulsant BH, Neufeld NH, Rothschild AJ, Voineskos AN, Whyte EM, Meyers BS; STOP-PD II Study Group. Predictors of relapse of psychotic depression: Findings from the STOP-PD II randomized clinical trial. J Psychiatr Res. 2023 Jan;157:285-290. doi: 10.1016/j.jpsychires.2022.12.011. Epub 2022 Dec 12. PMID 36535116
- [Derived] Voineskos AN, Mulsant BH, Dickie EW, Neufeld NH, Rothschild AJ, Whyte EM, Meyers BS, Alexopoulos GS, Hoptman MJ, Lerch JP, Flint AJ. Effects of Antipsychotic Medication on Brain Structure in Patients With Major Depressive Disorder and Psychotic Features: Neuroimaging Findings in the Context of a Randomized Placebo-Controlled Clinical Trial. JAMA Psychiatry. 2020 Jul 1;77(7):674-683. doi: 10.1001/jamapsychiatry.2020.0036. PMID 32101271
- [Derived] Flint AJ, Meyers BS, Rothschild AJ, Whyte EM, Alexopoulos GS, Rudorfer MV, Marino P, Banerjee S, Pollari CD, Wu Y, Voineskos AN, Mulsant BH; STOP-PD II Study Group. Effect of Continuing Olanzapine vs Placebo on Relapse Among Patients With Psychotic Depression in Remission: The STOP-PD II Randomized Clinical Trial. JAMA. 2019 Aug 20;322(7):622-631. doi: 10.1001/jama.2019.10517. PMID 31429896
- [Derived] Bingham KS, Whyte EM, Mulsant BH, Rothschild AJ, Rudorfer MV, Marino P, Banerjee S, Butters MA, Alexopoulos GS, Meyers BS, Flint AJ; STOP-PD Study Group. Health-related quality of life in remitted psychotic depression✰. J Affect Disord. 2019 Sep 1;256:373-379. doi: 10.1016/j.jad.2019.05.068. Epub 2019 May 28. PMID 31207561
- [Derived] Flint AJ, Meyers BS, Rothschild AJ, Whyte EM, Mulsant BH, Rudorfer MV, Marino P; STOP-PD II Study Group. Sustaining remission of psychotic depression: rationale, design and methodology of STOP-PD II. BMC Psychiatry. 2013 Jan 25;13:38. doi: 10.1186/1471-244X-13-38. PMID 23351522

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 269 participants were enrolled in the open-label phase. However, only 126 participants were eligible and consented to participate in the RCT phase. Reasons for not being eligible for the RCT phase included failure to achive remission criteria, discontinuation of treatment prior to the RCT, or decision by the participant not to consent to the RCT.
Period: Overall Study
Arm/Group | Sertraline + Olanzapine | Sertraline + Placebo
Started | 64 | 62
Completed | 43 | 24
Not Completed | 21 | 38
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 7 | 3
Not completed — Relapsed-all cause | 13 | 34
Not completed — Events not attributed to study meds | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sertraline + Olanzapine | Sertraline + Placebo | Total
Number analyzed (Participants) | 64 | 62 | 126
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 42 | 87
  >=65 years | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (15.1) | 55.7 (14.9) | 55.3 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 41 | 78
  Male | 27 | 21 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 15
  Not Hispanic or Latino | 58 | 53 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 9 | 15
  White | 54 | 49 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 23 | 47
  United States | 40 | 39 | 79
Hamilton Depression Rating Scale 17-Item Total Score [Mean (Standard Deviation); unit: units on a scale] — Hamilton Depression Rating Scale (HDRS) 17-item; The total score can range from 0-52. A higher score indicates worsening severity of depressive symptoms.
  units on a scale | 5.3 (3.6) | 5.6 (3.6) | 5.5 (3.6)
Weight [Mean (Standard Deviation); unit: pounds] | 178.6 (39.4) | 182.5 (39.8) | 180.5 (39.5)
Total Cholesterol level [Mean (Standard Deviation); unit: mg/dL] | 209.0 (51.3) | 220.4 (46.8) | 214.7 (49.3)
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] | 134 [90 to 186] | 121 [95 to 169] | 127 [95 to 180]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects at Risk of Relapse During the Randomized Phase.
Description: Relapse criteria include at least one of the following:
  1)Structured Clinical Interview for Diagnostic Statistical Manual #4 Trade Revision (DSM-IV-TR) Axis 1 Disorders (SCID) symptoms of major depression maintained over two weeks 2)17-item Hamilton Depression Rating Scale score of >17 maintained for more than one week + a mean increase of 5 points from entry into randomized phase 3)Re-emergence of psychosis for more than one week, with a SADS (Schedule for Affective Disorders and Schizophrenia) score of >2 on delusion or hallucination severity items 4)Significant clinical worsening defined as either emergence of high-risk of suicide, and/or development of mania for greater than one week, and/or psychiatric hospitalization.
Time Frame: From entry into randomized phase (baseline) and 36 weeks or earlier relapse
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline + Olanzapine | Sertraline + Placebo
Number analyzed (Participants) | 64 | 62
Participants | 13 | 34

2. Secondary Outcome: Changes in Metabolic Measures: Weight
Description: Change in weight from entry into randomized phase (baseline) and 36 weeks.
Time Frame: From entry into randomized phase (baseline) and 36 weeks
Measure: Mean (95% Confidence Interval); unit: pounds
Arm/Group | Sertraline + Olanzapine | Sertraline + Placebo
Number analyzed (Participants) | 64 | 62
pounds | 5.70 [3.30 to 8.11] | -3.11 [-5.41 to -0.81]

3. Secondary Outcome: Changes in Metabolic Measure: Cholesterol
Description: Change in cholesterol from entry into randomized phase (baseline) and 36 weeks.
Time Frame: From entry into randomized phase (baseline) and 36 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sertraline + Olanzapine | Sertraline + Placebo
Number analyzed (Participants) | 64 | 62
mg/dL | -0.46 [-14.90 to 5.57] | -22.28 [-32.71 to -11.86]

4. Secondary Outcome: Changes in Metabolic Measures: Triglycerides
Description: Change in triglycerides from entry into randomized phase (baseline) and 36 weeks.
Time Frame: From entry into randomized phase (baseline) and 36 weeks
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sertraline + Olanzapine | Sertraline + Placebo
Number analyzed (Participants) | 64 | 62
mg/dL | -3.85 [-31.68 to 23.99] | -18.18 [-30.05 to -6.31]

ADVERSE EVENTS:
Time Frame: 36 Weeks of RCT Phase
Description: Are based on items of the Udvalg for Kliniske Undersogelser Side effect scale (UKU), based on the following system: 1) Items with an increase of ≥2 points from baseline and items rated as a 3 on the UKU that were rated <3 at baseline. Exceptions include the following items: 35=Weight Gain, 36= Weight Loss. 2) Weight gain and weight loss AEs were determined by the following definitions: a. weight gain of >7% from pre-morbid weight, b. weight loss of >7% from pre-morbid weight in the RCT phase.
Arm/Group | Sertraline + Olanzapine | Sertraline + Placebo
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/62
Serious Adverse Events (participants affected / at risk) | 11/64 | 12/62
Other Adverse Events (participants affected / at risk) | 29/64 | 23/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline + Olanzapine (N=64) | Sertraline + Placebo (N=62)
Hospitalisation (Surgical and medical procedures) | 11 (11) | 12 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sertraline + Olanzapine (N=64) | Sertraline + Placebo (N=62)
Abnormal dreams (Psychiatric disorders) | 1 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (2)
Dizziness postural (Nervous system disorders) | 5 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Hypersomnia (Nervous system disorders) | 2 (2) | 3 (3)
Indifference (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4)
Libido decreased (Psychiatric disorders) | 4 (4) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (5)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 4 (5) | 2 (2)
Tension (Psychiatric disorders) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (5) | 3 (3)
Weight increased (Investigations) | 9 (11) | 3 (3)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/08/NCT01427608/Prot_SAP_000.pdf